CLINICAL TRIAL: NCT03372967
Title: Project IMPACT Immunizations (IMProving America's Communities Together) Scaled Demonstration
Status: Completed | Type: Observational
Sponsor: American Pharmacists Association Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 018
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Influenza
Keywords: preventable disease; vaccine; public health; vaccine history; point-of-care
MeSH Terms: conditions — Influenza, Human | interventions — Proto-Oncogene Proteins c-met; Patient Education as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comprehensive Vaccination History Review: Patients who receive a comprehensive vaccination history review at a participating pharmacy site will be eligible to: a) receive a vaccination forecast review, b) be evaluated for unmet vaccination needs, c) receive patient education, and d) have vaccination needs met.
  Interventions: Biological: Vaccine administration by a pharmacist; Behavioral: Unmet vaccination needs identified and met; Behavioral: Vaccination forecast review and patient education

INTERVENTIONS:
Biological: Vaccine administration by a pharmacist — Administration, number and types, of vaccines by a pharmacist
Behavioral: Unmet vaccination needs identified and met — Identification of unmet vaccination needs and having those needs met
Behavioral: Vaccination forecast review and patient education — Pharmacist review of the vaccination forecast and patient education on his/her vaccine needs

SUMMARY:
The primary objective of this study is to evaluate how implementing an innovative care model that provides the pharmacist access to a patient's vaccine history at the point-of-care impacts the pharmacist's ability to identify unmet vaccination needs and increase vaccination rates for routinely recommended adult vaccinations.

DETAILED DESCRIPTION:
This multi-site study will use a pre-post design with a population-based comparison group to investigate the impact of implementing an innovative care model on the pharmacist's ability to identify unmet vaccination needs and increase vaccination rates for routinely recommended adult vaccinations. The innovative care model enables the pharmacist to utilize a bi-directional IIS to assess patients' vaccination histories, identify unmet vaccination needs, and document the care provided. The project duration has been established to allow sufficient time for each pharmacy to implement the innovative care model and monitor each pharmacy for a 6-month study period. The American Pharmacists Association (APhA) Foundation has an a priori intent to publish the project results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible to be enrolled in the study include any person at least 18 years of age who is eligible for a comprehensive vaccination history review as determined by the pharmacist.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults eligible to receive vaccinations for preventable diseases
Sampling Method: Probability Sample
Enrollment: 6234 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Change in vaccination rates for routinely recommended adult vaccinations | 6 months
  Change from baseline rates

SECONDARY OUTCOMES:
Number of vaccines administered | 6 months
  Change from baseline rates
Types of vaccines administered | 6 months
  Change from baseline rates
Number of unmet vaccination needs that were identified and met | 6 months
  Measured through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Bluml, BPharm, Principal Investigator — American Pharmacists Association Foundation
Locations (22):
- United States (22):
  - Walmart Pharmacy, Atlantic, Iowa
  - Medicap Pharmacy, Carlisle, Iowa
  - NuCara Pharmacy, Coralville, Iowa
  - Eagle Pharmacy, Eagle Grove, Iowa
  - Medicap Pharmacy, Eldora, Iowa
  - Medicap Pharmacy, Indianola, Iowa
  - Towncrest Pharmacy, Iowa City, Iowa
  - Hy-Vee Pharmacy, Iowa City, Iowa
  - Walmart Pharmacy, Knoxville, Iowa
  - Osterhaus Pharmacy, Maquoketa, Iowa
  - Hy-Vee Pharmacy, Marion, Iowa
  - Walmart Pharmacy, Pella, Iowa
  - NuCara Pharmacy, Pleasant Hill, Iowa
  - NuCara Pharmacy, Traer, Iowa
  - Greenwood Pharmacy, Waterloo, Iowa
  - Meyer Pharmacy, Waverly, Iowa
  - Hy-Vee Pharmacy, West Des Moines, Iowa
  - NuCara Pharmacy, West Union, Iowa
  - Montross Pharmacy, Winterset, Iowa
  - Safeway Pharmacy, Bellevue, Washington
  - Safeway Pharmacy, Issaquah, Washington
  - Albertsons Sav-On Pharmacy, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No